CLINICAL TRIAL: NCT06734052
Title: Computer-guided Action Planning to Support Physical Activity (CAPPA) for Employees with Chronic Knee Symptoms
Acronym: CAPPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); Rush University (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Daniel Pinto, Associate Professor, Marquette University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR081007; 1R21AR081007-01A1 (NIH)
Record Dates: First submitted 2024-11-16; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis of Knee; Knee Pain Chronic
Keywords: knee symptoms; physical activity; Fitbit; accelerometer; Health coaching; remote coaching
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computer-guided Action Planning to support Physical Activity (CAPPA) (Experimental): Participants in the CAPPA Arm receive a Fitbit and health coaching using Computer-guided Action planning. Coaches will utilize the coaching software within www.myactionplans.com to guide the coaching interaction and support physical activity plan development. The emphasis is this arm is to create plans that are person-centered and driven by the participant. The action planning process is grounded in the conversational style of motivational interviewing and follows Brief Action Planning as a self-management support style. Coaches in the CAPPA arm will also have access to a custom Movement Dashboard which that uses Fitbit data to plot daily physical activity. The dashboard is coach-facing and is used to support coach dialogue about physical activity.
  There is scheduling flexibility: 4-12 visits over the 12-week period. Participants are strongly encouraged not to have a gap longer than three weeks between visits.
  Interventions: Behavioral: CAPPA
- Health education (Active Comparator): Participants in Arm 2 receive a Fitbit and health education delivered by a coach. Health education selects topics from the chronic disease self-management program that address common features of living with a chronic condition. Arm 2 avoids making specific plans and avoids discussion of physical activity. The emphasis in this arm is in providing education.
  There is scheduling flexibility, 4-12 visits over the 12-week period. Participants are strongly encouraged not to have a gap longer than three weeks between visits to keep the content fresh.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: CAPPA — See CAPPA arm description.
  Arms: Computer-guided Action Planning to support Physical Activity (CAPPA)
Behavioral: Health education — See health education arm description
  Arms: Health education

SUMMARY:
The goal of this clinical trial is to learn if a brief health coaching intervention based on an approach known as brief action planning + Fitbit can increase physical activity in employees with chronic knee symptoms who work for Advocate Aurora Health. The main questions it aims to answer are:

* Will a greater proportion of people in the health coaching intervention increase physical activity to at least 150 minutes of moderate-to-vigorous physical activity per week than a group of people with an attention-control intervention (Fitbit+health education coaching)?
* Can we predict who will not increase physical activity levels to at least 150 minutes of moderate-to-vigorous physical activity per week by the end of the study (3 and 6 months) based upon Fitbit data captured over the first four weeks?

Researchers will compare a health education coaching intervention + Fitbit to see if providing a Fitbit + attention control will increase physical activity to at least 150 minutes of moderate-to-vigorous physical activity per week among members of the attention-control group.

Participants will engage in

* Online study orientation and question and answer session
* Three assessment sessions (baseline, 3 months, 6 months)
* A 12 week intervention with no less than four (4) and no more than twelve (12) health coaching sessions. Physical activity health coaching will make action plans for health coaching. Health education coaching will focus on educating participants on non-physical activity factors related to a comprehensive management of chronic knee symptoms, such as managing fatigue, sleep hygiene, mindfulness, etc.

DETAILED DESCRIPTION:
Chronic knee symptoms (CKS) are associated with pain, loss of independence, and increased mortality. Rates of CKS are increasing, fueled by an aging, obese, and sedentary society. Because CKS first presents in working age adults, it is a major cause of work disability and work productivity loss.

Being physically active improves the health of adults who have ongoing (chronic) complaints of knee pain, knee stiffness, or challenges with moving around. Physical activity helps decrease pain, improve stiffness, and improve physical function as it relates to the knee. It also helps people improve their general health. Unfortunately, it is hard for many people to become more physically active. Physical activity can be inconvenient and uncomfortable for many people, and people who join physical activity programs often drop out of them after a short time (3-6 months). However, people are more likely to reach their physical activity goals if they work with a health coach who supports the process.

Health coaching often includes a combination of self-monitoring such as using smart devices to monitor outcomes plus the support of goal-directed behavior. Previous research has found that Fitbit tracking can improve behavior for some people who have CKS but not for others. Whereas we know people can receive benefit from coaching, the exact amount of coaching needed remains unknown. Discussion with employee stakeholders have informed our intervention desire as they have asked for a low resource form of coaching available through the workplace. The potential exists to support employees with CKS using an acceptable, low-resource coaching strategy.

The goal of this program is to test a brief, scalable PA coaching intervention that can assist employees with CKS attain and maintain healthy PA behavior in worksites in the Midwest. CAPPA is a 12-week pilot randomized controlled trial that will 1) use computer-guided action-planning behavioral intervention to support employees in making physical activity action plans for their health, 2) use data transmitted from a personal fitness tracker (Fitbit) to support coach and employee knowledge about PA performance, and 3) Inform on optimal step up times for participants who do not substantially increase PA. The CAPPA system will put PA feedback in a Movement Dashboard to support study participants. The CAPPA intervention will primarily use video chat to attain and sustain healthy PA behavior across worksites at Advocate Aurora Health.

Follow-up measures of PA, pain and physical function are planned at treatment completion and three months following study completion. Specific aims are to: 1) Estimate the efficacy of the intervention to increase objectively measured physical activity, 2) Examine the feasibility, acceptability and sustainability of the CAPPA intervention for the respective workplaces, and 3) Inform the initial step up time for future stepped interventions among participants not substantially increasing their physical activity. This study leverages the combined clinical and technologic expertise of the members of the Physical Activity in Rheumatology Research group at Northwestern University, Northwestern's Arthritis Center Accelerometer unit, Marquette University's Behavior, Engagement and Technology Assessment Lab and Ubiquitous Computing Lab, and Advocate Aurora Health.

This research could have a tremendous impact on improving symptoms and quality of life for those with CKS and early KOA. If treatments are successful at Advocate Aurora Health they may be employed in the services they provide to other organizations.

ELIGIBILITY:
Inclusion Criteria: Participants must be

1. Age >/= 18 years
2. Employed at a participating workplace
3. Report pain, aching or stiffness in or around the knee over the past 12 months
4. Report chronic pain, aching or stiffness in or around knee on most days for at least a month over the past 12 months
5. Have access to a device with active internet access to view study dashboard

Exclusion Criteria: Participants will be excluded if they

1. Currently meet CDC PA guidelines (per baseline accelerometer assessment)
2. Have had a joint replacement on the symptomatic side or plan to have one within the next year
3. Have serious medical conditions or impairments that, in the investigators' view, would create safety concerns in the trial such as uncontrolled hypertension (SPB>160 or diastolic ≥ 100 mm), or symptoms of unstable cardiac or pulmonary disease in the past month ( using the 2021 Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
4. Are unable to walk 50' with or without an assistive device
5. Plan to relocate from the region within the next year
6. Have limited English literacy
7. Carry a diagnosis of inflammatory arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of CDC-guideline based physical activity compliance | baseline, 3 month, 6month follow-up
  Proportion of people per treatment arm meeting CDC guidelines for aerobic physical activity. How many participants per group have achieved 150 minutes of weekly moderate-to-vigorous physical activity.

SECONDARY OUTCOMES:
Fitbit measured physical activity | baseline, week 1, week 2, week 3, week 4.
  Minutes of non-sedentary activity/day; Minutes of light, moderate-vigorous physical activity/day
Tampa Scale of Kinesiophobia | Baseline, 3 months, 6 months
  A self-report measure with 17 items used to measure fear of movement/(re)injury in chronic pain patients
Michigan Body Map | baseline, 3 month, 6 month follow-up
  The Michigan Body Map (MBM) is a self-report measure to assess body areas of chronic pain. The MBM can also quantify the degree of widespread body pain when assessing for centralized pain features.
Self-efficacy for physical activity | baseline, 3 month, 6 month follow-up
  This scale is a self-report of exercise self-efficacy.
Numeric Pain Rating Scale | baseline, 3 month, 6 month follow-up
  The NPRS is an 11-point scale scored from 0-10:
  1. "0" = no pain
  2. "10" = the most intense pain imaginable
WOMAC pain and physical function sub-scales | baseline, 3 month, and 6 month follow up
  The WOMAC subscales of pain (five questions), and physical function (17 questions). The subscale scores can vary, with pain ranging from 0 to 20 points; and physical function, 0 to 68 points. Higher scores represent worse pain and functional limitations.
PROMIS self reported outcomes | Baseline, 3 month, 6 month follow-up
  Computer-adaptive tests of self-reported physical function, pain interference, fatigue, and positive affect.
Performance-based outcomes - Timed up and Go | baseline, 3 month, 6 month follow-up
  Timed up and go - time it takes to stand from chair, walk 3 meters, return to chair and sit. measured in seconds
Performance-based outcomes - 4 meter walk | baseline, 3 month, 6 month follow-up
  Time it takes to walk four (4) meters. Measured in seconds
Performance-based outcomes - 5x sit-stand | baseline, 3 month, 6 month follow-up
  Time it takes to complete five (5) repetitions of the sit to stand movement. Timed from leaving the surface of the seat on the first sit-stand movement to contacting the seated surface on the fifth sit-stand movement.
Feasibility measure - recruitment rate | 3 month follow-up
  Number of participants engaging in screening process following targeted email or onset of recruitment campaigns.
Feasibility measures - consent rate | 3 month follow-up
  The proportion of eligible individuals who agreed to participate.
Feasibility measures - drop out rate | 3 month follow-up, 6 month follow-up
  Proportion of individuals who dropped out of the study at different stages of the study.
Feasibility measures - adherence to protocol | 3 month follow-up
  adherence to protocols - proportion of people who completed at least 4 coaching visits.
Feasibility measures - personnel retention | 3 month follow-up, 6 month follow-up
  number of personnel that left the study
Feasibility measures - fidelity | 3 month follow-up
  Proportion of reviewed coach recordings that followed prescribed coaching method.
Feasibility measures-qualitative | 3 month follow-up
  Qualitative sentiment regarding the ability of the coaching approach to integrate in an individual's work life.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pinto, PhD, Principal Investigator — Marquette University; Rowland W Chang, MD MPH, Principal Investigator — Northwestern University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available 1 year after NIH final report submission.
Access Criteria: IPD can be accessed by those who submit a proposal to the CAPPA leadership team describing planned analyses using a cloud-based online submission form. No formal data sharing agreement need be signed.
  To facilitate interpretation of the data, data dictionaries and protocols will be shared and associated with the relevant datasets via readme.txt files for the associated data.
  Data files will be archived using a SAS-based project-specific database with detailed documentation of any editing and data review adjudications while keeping original data files intact. Archived data files used to derive data analysis and original data files of non-identifiable, outcomes-related IPD will be shared.